CLINICAL TRIAL: NCT03704454
Title: The Use of Pycnogenol® to Alleviate Menopausal Symptoms Induced or Increased by Breast and Gynecological Cancer Treatments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Legacy Health System (Other)
Responsible Party: Principal Investigator, Reza Antoszewska, Legacy Health Foundation, Legacy Health System
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PYC001
Record Dates: First submitted 2018-10-04; First posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Climacteric; Menorrhagia, Menopausal; Menopause
MeSH Terms: conditions — Menorrhagia | interventions — pycnogenols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A - PYC & Placebo (Experimental): 50 mg of PYC for the first 4 weeks and then switch over to receive placebo for the following 4 weeks
  Interventions: Dietary Supplement: 50 mg PYC and then placebo
- Group B - PYC & Placebo (Experimental): 100 mg of PYC for the first 4 weeks and then switch over to receive placebo for the following 4 weeks
  Interventions: Dietary Supplement: 100 mg PYC and then placebo
- Group C - Placebo & PYC (Experimental): Placebo for the first 4 weeks and then switch over to 50 mg PYC for the following 4 weeks
  Interventions: Dietary Supplement: Placebo and then 50 mg PYC
- Group D - Placebo & PYC (Experimental): Placebo for the first 4 weeks and then switch over to 100mg PYC for the following 4 weeks
  Interventions: Dietary Supplement: Placebo and then 100 mg PYC

INTERVENTIONS:
Dietary Supplement: 50 mg PYC and then placebo — 4 weeks on PYC, then 4 weeks on placebo
  Arms: Group A - PYC & Placebo
Dietary Supplement: 100 mg PYC and then placebo — 4 weeks on PYC, then 4 weeks on placebo
  Arms: Group B - PYC & Placebo
Dietary Supplement: Placebo and then 50 mg PYC — 4 weeks on placebo, then 4 weeks on PYC
  Arms: Group C - Placebo & PYC
Dietary Supplement: Placebo and then 100 mg PYC — 4 weeks on placebo, then 4 weeks of PYC
  Arms: Group D - Placebo & PYC

SUMMARY:
This is a pilot study to test whether PYC can improve climacteric symptoms for women who have experienced either surgically or medically induced menopause as part of their treatment for breast or gynecologic cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patient currently is undergoing treatment for cancer
* Patient has menopausal symptoms induced either by surgical or medical (patient on tamoxifen or aromatase inhibitor) interventions for cancer
* > 18 years of age
* Willing to travel to a Legacy Health facility if necessary
* Agree to attend study visits outside of standard of care visits, if needed
* Willing to stop other supplements or medications that are aimed at treating menopausal symptoms at least 7 days before beginning study treatment
* Willing to engage in pre/post testing and survey/phone calls

Exclusion Criteria:

* Patient is currently undergoing chemotherapy treatment
* < 18 years of age
* Unable to comply with protocol
* Unable to provide written informed consent
* Investigator does not believe study participation is in the best interest of the patient
* Patient had concurrent menopausal symptoms prior to the start of cancer treatment
* Menopausal symptoms are unrelated to surgical or medical treatment of breast or gynecologic cancers

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-15 (Estimated); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
Menopause Rating Scale (MRS) | The MRS will be administered at baseline, after 4 weeks, after 8 weeks, 2 week follow-up (10 weeks), and 1 month follow up (12 weeks) with the intention of calculating DFB score at each time point.
  The MRS will be used to evaluate the efficacy of PYC in decreasing menopausal symptoms as compared to placebo. The difference-from-baseline (DFB) score will be calculated by taking the composite MRS score at 10 weeks and 12 weeks compared to the MRS score at baseline to determine whether or not PYC reduces symptoms, if the effects last beyond actively taking PYC, and if so, how long. The purpose of multiple time point assessments is two-fold: first, some patients will be taking placebo and some will be taking active drug in the first month, and vice versa during the second month. Therefore, an assessment needs to be done at each timepoint, weeks 4 and 8. Second, we are interested in understanding how long the symptoms management may last without actively taking drug, which accounts for the 10 week and 12 week timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Reza Antoszewska, NP-C, Principal Investigator — Legacy Health
Locations (3):
- United States (3):
  - Legacy Mt. Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Medical Center, Portland, Oregon
  - Legacy Meridian Park Medical Center, Tualatin, Oregon